CLINICAL TRIAL: NCT05053022
Title: A Study to Evaluate the Efficacy of Microneedling as a Stand-alone Treatment for Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crown Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-VL-21-04
Record Dates: First submitted 2021-08-26; First posted 2021-09-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: A proof of concept study to determine the safety and efficacy of Microneedling in patients with stable Vitiligo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microneedling with Skinpen Precision System (Experimental): Skinpen precision system will be used in accordance with the instructions in the IFU on the treatment area. A numbing cream will be applied at least 20-30 minutes before the Skinpen Precision system treatment is done. The affected areas will be treated at depths of up to 2.50mm. Treatment depth will be recorded for each treatment at every visit.
  Subjects will be dispensed with the Blue Lizard sunscreen and trained on proper use.
  Interventions: Device: Skinpen Precision System

INTERVENTIONS:
Device: Skinpen Precision System — Subjects will receive a total of 8-12 treatments with the Skinpen Precision system targeting their Vitiligo lesions.

SUMMARY:
This is a study that is being conducted in order to assess the efficacy of microneedling as a stand-alone treatment for vitiligo. Vitiligo is an autoimmune depigmentation disease of the skin that is characterized by the destruction of epidermal melanocytes by CD8+ T cells. The pathogenesis of Vitiligo has been linked to autoimmunity, oxidative stress, and genetic susceptibility.

DETAILED DESCRIPTION:
Microneedling is a minimally invasive technique developed for skin rejuvenation. In the treatment for vitiligo, the procedure causes micro-inflammations on the epidermis and enhances melanocytes and keratinocytes migration. This process leads to the stimulation and repigmentation of vitiligo areas. Several topical therapies such as Tacrolimus and 5-Fluorouracilused in conjunction with microneedling have yielded favorable repigmentation results. This study aims to evaluate the repigmentation rates of microneedled vitiligo patches without any topical medications other than sunscreen.

There will be a total of 8 -12 treatments over the course of 244 days, with subjects receiving a treatment every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, ages 18 through 60.
2. Clinical diagnosis of stable Vitiligo (no changes within the past 6 months) on any of the following body areas: face, neck, trunk, extremities, hands, feet (excluding digits).
3. Subjects in generally good health and free of any conditions which, in the opinion of the investigator, would interfere with the study assessments.
4. Subjects willing to discontinue all current therapies for vitiligo for the duration of the study.
5. Women of childbearing potential agree to take a urine pregnancy test at the Baseline visit and Final visit.
6. Individuals that are willing to provide written informed consent and are able to read, speak, write and understand the informed consent document.
7. Willingness to cooperate and participate by following study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.

Exclusion Criteria:

1. Individuals diagnosed with known allergies to facial or general skin care products.
2. Individuals who have presence of an active systemic or local skin disease, apart from vitiligo, that may affect wound healing. Uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
3. Individuals with sensitivity to topical lidocaine, stainless steel, nickel, or chromium
4. Individuals who have a recent or current history of inflammatory skin disease or cancerous/pre-cancerous lesion.
5. Subjects currently or within the past 3 months on Vitiligo topical or systemic treatments.
6. Use of skin lighteners or bleaching agents; hydroquinone, phenol peels or harsh chemicals.
7. Individuals who have the inability to understand instructions or to give informed consent.
8. Individuals who have a history of chronic drug or alcohol abuse.
9. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
10. Individuals who are current smokers.
11. Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
12. Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
13. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
14. Individuals who are currently participating in any other study involving the use of investigational device or drugs at another research facility or doctor's office within 4 weeks prior to inclusion into the study.
15. Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other facial cosmetic treatments; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment (PGA) | Through Study Completion, over the course of 244 days
  PGA to be completed starting at Visit 2 and on, prior to each treatment. The primary endpoint is to achieve Grade 2, 3 or 4 on the PGA Scale comparing photographs from baseline to visits 12, 13, and 14.
  This is a 5 Grade Repigmentation Scale. This assessment uses a scale of G0-G4. This global assessment will be done by the investigator starting at Visit 2 and afterwards.
  G4 Excellent > 75% Repigmentation G3 Very Good 50%-75% Repigmentation G2 Good 25%-50% Repigmentation G1 Satisfactory <25% Repigmentation G0 Poor No Repigmentation

SECONDARY OUTCOMES:
Subject's assessment of their pre and post-treatment images using the Vitiligo Noticeability Scale (VNS) | Through Study Completion, over the course of 244 days
  Subject's assessment of their pre and post-treatment images using the Vitiligo Noticeability Scale. A score of 3,4, or 5 indicates the success of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Crown Laboratories, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No